CLINICAL TRIAL: NCT04179539
Title: Gallium68 Ventilation/Perfusion PET/CT for Pulmonary Embolism Diagnosis: a Diagnostic Accuracy Study vs CT Pulmonary Angiography
Brief Title: Ga68 V/Q PET/CT for Pulmonary Embolism Diagnosis: a Diagnostic Accuracy Study vs CT Pulmonary Angiography
Acronym: PETEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETEP (29BRC18.0275); 2018-004723-36 (EudraCT Number)
Record Dates: First submitted 2019-11-12; First posted 2019-11-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients with suspected acute PE undergo CTPA and V/Q PET/CT imaging within 24 hours. V/Q PET/CT images are not used for patients management.
  After completion of inclusion, central readings will be independently conducted:
  * CTPA will be interpreted by two radiologists, blinded to the results of any clinical information or imaging test results. The results of this interpretation will be used as a reference standard.
  * V/Q PET/CT will be interpreted by two independant nuclear medicine physicians, blinded to the results of any clinical information or imaging test results (including the reference standard).
  Interventions: Diagnostic Test: V/Q PET/CT; Diagnostic Test: CTPA

INTERVENTIONS:
Diagnostic Test: V/Q PET/CT — Ventilation images are acquired after inhalation of Galligas prepared using a Technegas generator (Cyclopharm, Sydney, Australia). The patients is placed in a supine position and inhaled Galligas using the standard ventilation technique. Ventilation images are then acquired. Without the patient moving, 68Ga-MAA are then injected. Perfusion PET images are then acquired
Diagnostic Test: CTPA — CTPA will be done according to the usual protocol in the radiology department of the investigator center

SUMMARY:
This study evaluates the diagnostic accuracy (sensitivity, specificity) of V/Q PET/CT for the diagnosis of pulmonary embolism (PE), using CT pulmonary angiography as a reference standard.

DETAILED DESCRIPTION:
V/Q PET/CT imaging is now possible by substituting 99mTc with 68Ga, a positron-emitting radionuclide, using the same carrier molecules as conventional V/Q imaging. Ventilation imaging can be performed with 68Ga-carbon nanoparticles using the same synthesis device as Technegas. Perfusion imaging can be performed with 68Ga-macroaggregated albumin (68Ga-MAA).Technical advantages of PET compared to SPECT include higher sensitivity, higher spatial and temporal resolution and superior quantitative capability. This offers the opportunity to improve the accuracy of V/Q imaging in patients with suspected PE, while decreasing the acquisition time.

The aim is to perform a formal diagnostic accuracy study of V/Q PET/CT for PE, using CTPA as a reference standard.

Patients with suspected acute PE undergo CTPA and V/Q PET/CT imaging within 24 hours.

V/Q PET/CT images are not used for patients management.

After completion of inclusion, central readings of scans will be conducted independently.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected first episode of acute PE,
* Age ≥ 18 years .
* Insured patient.

Exclusion Criteria:

* Patients with a clinically suspected massive PE.
* Contraindication to contrast media (including renal insufficiency with creatinine clearance < 30 ml/min).
* Inability to perform CTPA and V/Q PET/CT within 24 hours.
* History of deep vein thrombosis or PE
* Unable/unwilling to give informed consent.
* Pregnancy / breast-feeding.
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of V/Q PET/CT for PE diagnosis | Baseline
  Proportion of patients with a positive V/Q PET/CT among patients with PE according to the reference standard (CTPA).
Specificity of V/Q PET/CT for PE diagnosis | Baseline
  Proportion of patients with a negative V/Q PET/CT among patients without PE according to the reference standard (CTPA).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de BREST, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Blanc-Beguin F, Elies P, Robin P, Tripier R, Kervarec N, Lemarie CA, Hennebicq S, Tromeur C, Cogulet V, Salaun PY, Le Roux PY. 68Ga-Labelled Carbon Nanoparticles for Ventilation PET/CT Imaging: Physical Properties Study and Comparison with Technegas(R). Mol Imaging Biol. 2021 Feb;23(1):62-69. doi: 10.1007/s11307-020-01532-6. Epub 2020 Sep 4. PMID 32886302